CLINICAL TRIAL: NCT02722187
Title: The Role of Microsurgery in Surgical Treatment of Varicocele.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: microvl/2015
Record Dates: First submitted 2016-03-24; First posted 2016-03-29 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Varicocele; Infertility
MeSH Terms: conditions — Varicocele; Infertility

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- microsurgery (Experimental): 40 patients will undergo subinguinal microscopic varicocelectomy
  Interventions: Procedure: subinguinal microscopic varicocelectomy
- laparoscopy (Active Comparator): 20 patients will undergo laparoscopic varicocelectomy
  Interventions: Procedure: laparoscopic varicocelectomy

INTERVENTIONS:
Procedure: subinguinal microscopic varicocelectomy
  Arms: microsurgery
Procedure: laparoscopic varicocelectomy
  Arms: laparoscopy

SUMMARY:
This study is to set the place of microsurgery in surgical treatment od varicocele in infertile male. Fourty patients will undergo microsurgical subinguinal varicocelectomy while the control group consisting of 20 patients wil undergo laparoscopic varicocelectomy.

ELIGIBILITY:
Inclusion Criteria:

* clinical varicocele
* infertility duration of min one year
* poor semen quality
* otherwise unexplained infertility in the couple

Exclusion Criteria:

* female infertility

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate after the intervention | one yaer after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Chair and Department of Urology Warsaw Medical University., Warsaw, Poland

REFERENCES:
- [Result] Diegidio P, Jhaveri JK, Ghannam S, Pinkhasov R, Shabsigh R, Fisch H. Review of current varicocelectomy techniques and their outcomes. BJU Int. 2011 Oct;108(7):1157-72. doi: 10.1111/j.1464-410X.2010.09959.x. Epub 2011 Mar 24. PMID 21435155
- [Result] Ollandini G, Liguori G, Ziaran S, Malek T, Mazzon G, de Concilio B, Bucci S, Benvenuto S, Belgrano E, Trombetta C. Varicocele treatment: a 2-centers comparison between non microsurgical open correction, laparoscopic approach and retrograde percutaneous sclerotization on 463 cases. Arch Ital Urol Androl. 2013 Sep 26;85(3):143-8. doi: 10.4081/aiua.2013.3.143. PMID 24085237
- [Result] Abdel-Meguid TA, Al-Sayyad A, Tayib A, Farsi HM. Does varicocele repair improve male infertility? An evidence-based perspective from a randomized, controlled trial. Eur Urol. 2011 Mar;59(3):455-61. doi: 10.1016/j.eururo.2010.12.008. Epub 2010 Dec 21. PMID 21196073
- [Result] Cayan S, Shavakhabov S, Kadioglu A. Treatment of palpable varicocele in infertile men: a meta-analysis to define the best technique. J Androl. 2009 Jan-Feb;30(1):33-40. doi: 10.2164/jandrol.108.005967. Epub 2008 Sep 4. PMID 18772487
- [Result] Al-Kandari AM, Shabaan H, Ibrahim HM, Elshebiny YH, Shokeir AA. Comparison of outcomes of different varicocelectomy techniques: open inguinal, laparoscopic, and subinguinal microscopic varicocelectomy: a randomized clinical trial. Urology. 2007 Mar;69(3):417-20. doi: 10.1016/j.urology.2007.01.057. PMID 17382134
- [Result] Watanabe M, Nagai A, Kusumi N, Tsuboi H, Nasu Y, Kumon H. Minimal invasiveness and effectivity of subinguinal microscopic varicocelectomy: a comparative study with retroperitoneal high and laparoscopic approaches. Int J Urol. 2005 Oct;12(10):892-8. doi: 10.1111/j.1442-2042.2005.01142.x. PMID 16323983